CLINICAL TRIAL: NCT05089370
Title: Oral Decitabine/Cedazuridine (DEC-C) in Combination With Nivolumab as a Strategy to Enhance the Efficacy of Immune Checkpoint Blockade in Unresectable or Metastatic Mucosal Melanoma
Brief Title: Oral Decitabine/Cedazuridine (DEC-C) in Combination With Nivolumab for Patients With Mucosal Melanoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Comprehensive Cancer Network (Network); Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-3518.cc; NCI-2021-10828 (Other: CTRP); 2021-IST-DECC-000076 (Other: NCCN)
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Decitabine; cedazuridine; decitabine and cedazuridine drug combination; Nivolumab

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-arm trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Decitabine/Cedazuridine (DEC-C) and Nivolumab in Mucosal Melanoma (Experimental)
  Interventions: Combination Product: Oral Decitabine/Cedazuridine (DEC-C) in Combination with Nivolumab

INTERVENTIONS:
Combination Product: Oral Decitabine/Cedazuridine (DEC-C) in Combination with Nivolumab — Activation of the RIG-I innate immune pathway and increased expression of tumor antigens and pro-immune genes during Nivolumab treatment may enhance the frequency and activity of anti-tumor immune cells (CD4+ and CD8+ T-cells, NK cells) and reduce the frequency and activity of immunosuppressive cells (MDSCs, Tregs) (1-4), increasing the overall effectiveness and success of Nivolumab treatment. This pilot clinical trial will demonstrate whether combinatorial immunotherapeutic approaches that target epigenetic immune repression and RIG-I activity can favorably alter the tumor immune cell microenvironment and benefit mucosal melanoma patients.

SUMMARY:
Activation of the RIG-I innate immune pathway and increased expression of tumor antigens and pro-immune genes by DEC-C during Nivolumab treatment may enhance the frequency and activity of anti-tumor immune cells (CD4+ and CD8+ T-cells, NK cells) and reduce the frequency and activity of immunosuppressive cells. This may increase the overall effectiveness and success of Nivolumab treatment. This pilot clinical trial will demonstrate whether combinatorial immunotherapeutic approaches that target epigenetic immune repression and RIG-I activity can favorably alter the tumor immune cell microenvironment and benefit patients with mucosal melanoma.

DETAILED DESCRIPTION:
This is a Phase Ib/II investigator-initiated open label trial of the combination of DEC-C and Nivolumab treatment.

This is a single-center study to be conducted at the University of Colorado Cancer Center (UCHealth central campus). A complete and current listing of investigators, research personnel, and research facilities participating in this study will be maintained throughout the duration of this study on applicable study required forms such as an FDA Form 1572, the COMIRB Research Personnel Form, and/or a UCCC Protocol Contact List, incorporated herein by reference.

Phase Ib: A time-to-event Bayesian optimal interval (TITE-BOIN) design will be used to assess the RP2D during phase 1b. The BOIN design is a model assistant approach used in phase I clinical trials for finding the maximum tolerated dose (MTD). The Investigator anticipates a maximum of 9 patients treated at the RP2D in Phase 1b dose de-escalation and considers as subjects in stage 1 of phase 2.

Phase II: The objective of Phase II is to preliminarily evaluate the efficacy and further evaluate safety of the combination at the RP2D. The phase II cohort will enroll patients using the established RP2D of DEC-C from the phase Ib portion in combination with standard doses of Nivolumab. Patients treated at the RP2D in Phase 1b will be included in analysis for the Phase II component of this study. All patients enrolled at the RP2D level and receiving any DEC-C treatment will be included in the efficacy and safety/tolerability endpoint analysis. The results indicate that the objective response rate (ORR) to anti-PD1 in mucosal melanoma patients at our institution is 20%. The Investigator hypothesizes ORR for the combination will be 43%, a 23% absolute improvement over the anti-PD1 treatment. Simon's 2-stage design will be used to evaluate the ORRs. The null hypothesis that the ORR is 20% will be rejected if there are 3 or more responses among the 11 patients (including phase Ib RP2D patients). The design yields a type I error rate of 001 and power of 80% when the true response rate is 43%. The total sample size required for the Phase II will depend on the number of patients treated at the RP2D during Phase 1b, and it is estimated the total sample size will be in the range of 19-21 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be a male or female aged 18-100.
4. Histologically confirmed diagnosis of advanced mucosal melanoma (unresectable Stage III or Stage IV Melanoma). Anatomical locations for primary site of mucosal melanoma include oral cavity (excluding lip), nasopharynx, vagina/vulva, and rectum.
5. Prior immune checkpoint blockade therapy, including anti-PD1 and anti-CTLA4 for unresectable locally advanced or metastatic disease, is allowed. The combination of anti-PD1 and anti-CTLA4 is also allowed as a prior line of therapy. Study therapy must be initiated within 30 days of previous immune checkpoint blockade therapy (excluding adjuvant anti-PD1 and anti-CTLA4).
6. Patients must have systemic cross-sectional imaging (PET/CT or CT of chest, abdomen, and pelvis) with radiographically measurable, by immune-RECIST (RECIST) criteria, or clinically measurable disease.
7. Previously treated brain metastatic disease is allowed. Stability of brain metastases must be confirmed by MRI > 4 weeks from most recent treatment and within 4 weeks of initiating study therapy.
8. Patients must have an ECOG performance status of 0 or 1 (Table 5).
9. Patients must have adequate bone marrow function as evidenced by all of the following: ANC ≥ 2,500 microliter (mcL); platelets ≥ 100,000/mcL; Hemoglobin ≥ 10 g/dL.
10. Patients must have adequate hepatic function as evidenced by the following: total bilirubin ≤ 1.5 x institutional upper limit of normal (IULN) (except Gilbert's Syndrome, who must have a total bilirubin < 3.0 mg/dL), and SGOT (AST) and SGPT (ALT) and alkaline phosphatase ≤ 2.5 x ULN.
11. Patients must have adequate renal function as evidenced by ONE of the following: serum creatinine ≤ 2.0 x ULN OR measured or calculated creatinine clearance ≥ 40 mL/min.
12. Patients known to be HIV positive are eligible if they meet the following criteria within 30 days prior to registration: stable and adequate CD4 counts (≥ 350 mm3), and serum HIV viral load of < 25,000 IU/ml. Patients may be on or off anti-viral therapy so long as they meet the CD4 count criteria.
13. Women of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. Women/men of reproductive potential must have agreed to use an effective contraceptive method for the course of the study through 120 days after the last dose of study medication. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. A woman is considered to be of "reproductive potential" as defined in section 5.3.2.
14. Patients must be willing to have archived tumor specimens utilized for correlative studies if available.
15. Patients must consent to have biopsies performed prior to treatment and around cycle 2 during study. However, in the event that tumor is inaccessible, the biopsy is not in the subject's best interest, or the patient refuses biopsy during course of the study, patients will be allowed to remain on study.

Exclusion Criteria:

1. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, lobular carcinoma of the breast in situ, atypical melanocytic hyperplasia or melanoma in situ, treated and stable thyroid cancer, adequately treated Stage I cancer (including multiple primary melanomas) from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for three years.
2. Patients must not currently be on other drugs metabolized by CDA.
3. Prior cytotoxic chemotherapy treatment received within 30 days of study enrollment.
4. Patients with leptomeningeal disease.
5. Current immunosuppressive therapy including >10mg/day of prednisone within 14 days of enrollment is not permitted. Inhaled or topical steroids, and adrenal replacement steroid doses ≤10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
6. Patients must not have known active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection prior to registration.
7. Patients must not have active autoimmune disease that has required systemic treatment in past 2 years from date of enrollment (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
8. Patients must not have a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
9. Patients must not have received live vaccines within 42 days prior to enrollment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, shingles, yellow fever, rabies, BCG, and typhoid (oral) vaccine. Seasonal influenza and COVID-19 vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
10. Patients must not have a history or current evidence of any condition, therapy or laboratory abnormality that might confound the trial results, interfere with the patient's participation for the full duration of the trial, or indicate that participation in the trial is not in the patient's best interests, in the opinion of the treating investigator.
11. Patients must not be pregnant or lactating.
12. Treatment with any investigational agent within 30 days of first administration of study treatment is not permitted.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Determine the safety of DEC-C in combination with Nivolumab unresectable, locally advanced, or metastatic mucosal melanoma patients. | 24 months
  Determine the safety and tolerability of DEC-C in combination with Nivolumab by evaluating adverse events (AEs) using CTCAEv5.0 criteria and establishing the recommended phase 2 dose (RP2D) of DEC-C.

SECONDARY OUTCOMES:
Determine the response rate to DEC-C in combination with Nivolumab in unresectable, locally advanced, or metastatic mucosal melanoma patients | 24 months
  Evaluate the rate of subjects that achieve an objective response (ORR) to DEC-C in combination with Nivolumab by radiographic assessment using iRECIST criteria.
Determine if the addition of DEC-C to Nivolumab increases progression free survival (PFS) and overall survival (OS) in unresectable, locally advanced, or metastatic mucosal melanoma patients. | 24 months
  Evaluate and estimate progression free survival (PFS) and overall survival (OS) in unresectable locally advanced and metastatic mucosal melanoma patients at 24 months post-study.

OTHER OUTCOMES:
Evaluate the effect of DEC-C in combination with Nivolumab on circulating and tumor immune cell profiles. | 24 months
  Compare the frequency and activity of circulating and tumor immune cells pre- and on- treatment by flow cytometry.
Determine the effect of DEC-C in combination with Nivolumab on global hypomethylation and RIG-I pathway gene expression in circulating cells and tumor cells. | 24 months
  Evaluate pre- and on- treatment levels of global hypomethylation and RIG-I pathway gene expression in circulating and tumor cells by qRT-PCR.
Determine the effect of DEC-C in combination with Nivolumab on circulating and tumor innate immune sensing cytokines and proteins. | 24 months
  Analyze pre- and on- treatment levels of circulating and tumor immune cytokines and proteins by Olink proteomics analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Martin McCarter, Principal Investigator — Colorado Research Center
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with the NCCN per research agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: within one year of enrollment completion.
Access Criteria: de-identified data